CLINICAL TRIAL: NCT05771129
Title: Feasibility and Safety Evaluation of the Pulsed Electric Field Ablation System on Patients With Chronic Bronchitis
Brief Title: Feasibility Study of the Pulsed Electric Field Ablation System in Treating Chronic Bronchitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiayuan Sun (Other)
Collaborators: Zhouling (Shanghai) Medical Appliance Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Jiayuan Sun, Director, Department of Endoscopy, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS22097
Record Dates: First submitted 2023-02-22; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Chronic Bronchitis
Keywords: Chronic Bronchitis; Chronic Obstructive Pulmonary Disease; Pulsed Electric Field Ablation; Safety Evaluation; Feasibility Study
MeSH Terms: conditions — Bronchitis, Chronic; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulsed Electric Field Ablation System was used in treating chronic bronchitis (Experimental): All participants meet inclusion and exclusion criteria and signed the ICF will be enrolled to experimental arm.
  Interventions: Device: Pulse electric field ablation system developed by Zhouling (Shanghai) Medical Appliance Co., Ltd.

INTERVENTIONS:
Device: Pulse electric field ablation system developed by Zhouling (Shanghai) Medical Appliance Co., Ltd. — Pulsed electric field ablation instrument is a therapeutic instrument based on the irreversible electroporation (IRE) mechanism. The high frequency short duration energy is delivered via a disposable pulse ablation catheter through the bronchoscope and act on the bronchial mucosa, through which goblet cell hyperplasia and airway mucus secretion will be alleviated. The entire treatment consists of two procedure sessions that will be performed one month apart. The first treatment procedure consists of a baseline biopsy of the airway mucosa followed by the treatment of the right lung. The second procedure consists of a biopsy of the treated airway, followed by the left-side treatment. A third bronchoscopy will be performed three months following the first treatment and mucosa-biopsy will be conducted to evaluate the histopathological change in mucus producing cells after treatment. Subjects will also be required to fill questionnaire and complete several examinations during follow-up.

SUMMARY:
To preliminarily evaluate the safety and feasibility of the pulsed electric field ablation system independently developed by Zhouling (Shanghai) Medical Appliance Co., Ltd. in the treatment of chronic bronchitis.

DETAILED DESCRIPTION:
Pulsed electric field ablation instrument is a therapeutic instrument based on the irreversible electroporation (IRE) mechanism. The high frequency short duration energy is delivered via a disposable pulse ablation catheter through the bronchoscope and act on the bronchial mucosa, through which goblet cell hyperplasia and airway mucus secretion will be alleviated.

The entire treatment consists of two procedure sessions that will be performed one month apart. The first treatment procedure consists of a baseline biopsy of the airway mucosa followed by the treatment of the right lung. The second procedure (one month after right-sided lung treatment) consists of a biopsy of the treated airway, followed by the treatment of the left lung. All procedures will be performed under general anaesthesia. Treatment is considered complete once the two bronchoscopic ablation procedures are successfully completed.

A third bronchoscopy will be performed three months following the first treatment where mucosa-biopsy will be taken from the previously treated airway sites to evaluate the histopathological evidence of change in mucus producing cells within the airway after treatment. Subjects will be required to fill questionnaire (SGRQ and CAT ) and complete several examinations (including chest CT scans, respiratory function tests, etc.) during follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subject's age is ≥35 years and ≤80 years;
2. Subject has chronic bronchitis, defined as productive cough for at least three months in each of two successive years, whereas other causes of productive cough have been ruled out.
3. Subject has a CAT score ≥ 10.
4. Subject has a SGRQ score ≥ 25.
5. Subject's responses to the first two questions of the CAT questionnaire sum to ≥ 7 points or the sum is 6 points and the subject's total CAT score is > 20 points.
6. Subject has post -bronchodilator FEV1/FVC < 0.7.
7. Subject has post-bronchodilator FEV1 percent predicted of ≥ 30%.
8. Subject is receiving guideline directed pharmacotherapy which includes one or more long-acting bronchodilator (LAMA, LABA) with or without an inhaled corticosteroid for at least 8 weeks prior to randomization, unless the patient has attempted such therapy within the past 1 year without significant clinical response or had an adverse reaction.
9. Subject has a cigarette smoking history of at least ten pack years, and has had quit smoking for at least 6 months before enrollment (cigarettes, e-cigarettes, etc.), and agreed to remain non-smoking during the study;
10. In the opinion of the investigator, subject is able to undergo 3 bronchoscopies under general anesthesia (including mucosal biopsy), is willing to participate in the study, and is able to follow the study follow-up plan.

Exclusion Criteria:

1. Subject has known unresolved lower respiratory tract infection (e.g., pneumonia, mycobacterium avium-intracellulare infection (MAI), fungus, tuberculosis, etc).
2. Subject has a steroid-dependent condition requiring >10 mg of oral corticosteroid per day.
3. Subject has any implantable electronic device (e.g., pacemaker, cardioverter defibrillator) that cannot be turned off during the procedure.
4. Subject has a history of ventricular tachy-arrhythmia or clinically significant atrial tachyarrhythmia within the past two years, unless the arrhythmia has been treated and/or patient is in regular rhythm during the screening phase.
5. Subject has unresolved lung cancer.
6. Subject has a pulmonary nodule or cavity that in the judgement of the investigator may require intervention during the course of the study.
7. Subject had prior lung surgery, such as lung transplant, LVRS, lobectomy, lung implant/prosthesis, metal airway stent, valves, coils or bullectomy, etc. Previous sub-lobectomy, previous history of pneumothorax but no pneumonectomy, previous pleural disease but no surgical intervention are not the exclusion criteria;
8. Subject has emphysema of greater than or equal to 50% as quantified on baseline HRCT scan (low attenuation area less than -950HU) as determined by the CT.
9. Subjects had a history of asthma diagnosed at an age < 30.
10. Subject has clinically significant bronchiectasis which clinical symptoms of cough and phlegm affect the subject's quality of life.
11. BMI<18 or > 35;
12. Subject has a serious medical condition that, in the investigator's opinion, could endanger the patient's life or compromise patient safety or confound the interpretation of the patient's response to therapy (e.g., congestive heart failure, cardiomyopathy, or myocardial infarction in the past year, renal failure, liver disease cerebrovascular accident within the past 6 months, uncontrolled diabetes (HbA1c >8%), uncontrolled hypertension (diastolic BP >100mmHg) or autoimmune disease requiring treatment with immunosuppressant medications or a disease requiring chemotherapy).
13. Subject has uncontrolled GERD.
14. Subjects are known to have contraindications for bronchoscopy or general anesthesia, or to be allergic to related medications (i.e., lidocaine, atropine, benzodiazepines) and unable to respond to medications.
15. Subject is pregnant, nursing, or planning to get pregnant during study duration.
16. Subject is currently participating in another clinical study involving an investigational product (with interventional measures).

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-03-10 (Estimated); Primary Completion 2024-03-10 (Estimated); Study Completion 2025-03-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate the rate of adverse events and severe adverse events associated with pulsed electric field ablation systems | Within 30 days after either the first or second study procedure
  1. Index Name: Incidence of surgical or device-related adverse events during and within 1 month of bilateral lung ablation Observation purpose: To evaluate the safety of pulsed electric field ablation. Definition of index: To evaluate the adverse events according to CTCAE v5.0 and evaluate its correlation with the device itself or the operation and calculate the incidence rate of serious adverse events related to the device and the operation treatment.
  2. Index Name: The incidence of surgery-or device-related serious adverse events. Observation purpose: To evaluate the safety of pulsed electric field ablation. Definition of index: To evaluate the serious adverse events according to CTCAE v5.0 and evaluate its correlation with the device itself or the operation and calculate the incidence rate of serious adverse events related to the device and the operation treatment.

SECONDARY OUTCOMES:
Improvements in COPD Version of the St. George Respiratory Questionnaire (SGRQ-C) | 6 and 12 months after bilateral treatment
  To evaluate the changes from baseline in the total score of the COPD Version of the St. George Respiratory Questionnaire (SGRQ-C) at 6 and 12 months after bilateral surgery.
Improvements in COPD Assessment Test (CAT) score | 6 and 12 months after bilateral treatment
  To evaluate changes from baseline in the COPD Assessment Test (CAT) score at 6 and 12 months after bilateral surgery.
Clinical Efficacy - Pulmonary Function | 6 and 12 months after bilateral treatment
  To evaluate changes from baseline in forced expiratory volume in the first second (FEV1) in pulmonary function tests (PFT) at 6 and 12 months after bilateral surgery.
Pathological examination-goblet cell proliferation score | 3 months after treatment on the right side
  Baseline, 1 month and 3 months after surgery, the mucosa of the right airway should be biopsied, and obtained tissue should be stained with HE and PAS, in which the proliferation of goblet cells should be compared and scored (semi-quantitative , goblet cells: ciliated cells: 0 point, normal, 1: 10; 1 point, mild hyperplasia, 1: 3-10; 2 points, moderate hyperplasia, 1: 1; 3 points, severe hyperplasia, > 1: 1)
Acute exacerbation | 12 months after bilateral treatment
  To evaluate the times of moderate and severe acute exacerbation and the length of hospitalization within 12 months after bilateral operation.
  Acute exacerbation is defined as the simultaneous occurrence of two or more exacerbations or new episodes of respiratory symptoms, such as short of breath, cough, expectoration, dyspnea or chest tightness, and at least one respiratory symptom lasts for three days or more, resulting in the need for short-acting bronchodilators, or the use of antibiotics and/or oral glucocorticoids (moderate acute exacerbation), or the need for hospitalization or emergency treatment (severe acute exacerbation)
Distal Airway Volume | 6 and 12 months after bilateral treatment
  To evaluate changes from baseline in distal Airway Volume (based on expiratory phase HRCT imaging analysis) at 6 and 12 months after bilateral surgery.
Incidence of device defects | After bilateral treatment, assessed up to 2 months
  It refers to the unreasonable risks that may endanger human health and life safety in the normal use of medical devices during the clinical trials, such as labeling errors, quality problems, failures, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, MD., PhD., Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hartman JE, Garner JL, Shah PL, Slebos DJ. New bronchoscopic treatment modalities for patients with chronic bronchitis. Eur Respir Rev. 2021 Jan 19;30(159):200281. doi: 10.1183/16000617.0281-2020. Print 2021 Mar 31. PMID 33472961
- [Background] Herth FJF, Kontogianni K, Brock J. Endoscopic Options for Moderate COPD, Chronic Bronchitis, and Uncontrolled Asthma. Semin Respir Crit Care Med. 2022 Aug;43(4):552-558. doi: 10.1055/s-0042-1747939. Epub 2022 Jun 1. PMID 35649430
- [Background] Valipour A, Fernandez-Bussy S, Ing AJ, Steinfort DP, Snell GI, Williamson JP, Saghaie T, Irving LB, Dabscheck EJ, Krimsky WS, Waldstreicher J. Bronchial Rheoplasty for Treatment of Chronic Bronchitis. Twelve-Month Results from a Multicenter Clinical Trial. Am J Respir Crit Care Med. 2020 Sep 1;202(5):681-689. doi: 10.1164/rccm.201908-1546OC. PMID 32407638